CLINICAL TRIAL: NCT05398341
Title: A Prospective Cohort Post Market Registry Evaluating Outcomes of Bridge-Enhanced ACL Restoration (BEAR®)
Status: Active, not recruiting | Type: Observational
Sponsor: Miach Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: Bridge Registry
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; ACL surgery; ACL tear; Torn ACL; BEAR Implant; BEAR ACL; BEAR restoration; Bridge-enhanced ACL restoration; ACL restoration; ACL implant bridge
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Cohort: There will be a prospective cohort for all subjects scheduled to undergo ACL surgery with the BEAR Implant that are willing to provide consent.
  Interventions: Device: The BEAR® Implant
- Retrospective Cohort: A retrospective cohort will be available for all subjects treated with the BEAR Implant at each participating site. There is no control group.
  Interventions: Device: The BEAR® Implant

INTERVENTIONS:
Device: The BEAR® Implant — The BEAR Implant is a bovine collagen-based implant. The bovine tissue is sourced from countries that are free of bovine spongiform encephalopathy [BSE] and is further treated to remove bovine cell fragments and DNA.
  The BEAR® (Bridge Enhanced ACL Restoration) Implant is a bovine extracellular matrix collagen-based implant for treatment of anterior cruciate ligament (ACL) injuries. The BEAR® Implant is indicated for skeletally mature subjects at least 14 years of age with a complete rupture of the ACL. Subjects must have an ACL stump attached to the tibia to construct the repair.

SUMMARY:
The purpose of the Bridge Registry is to assess real-world performance of the FDA approved BEAR Implant.

DETAILED DESCRIPTION:
This is an observational study, where the BEAR Implant will be evaluated in a real-world setting. The registry seeks to enroll consecutive uses of the BEAR Implant at participating sites. There will be a prospective cohort for all subjects scheduled to undergo ACL surgery with the BEAR Implant that are willing to provide consent. A retrospective cohort will be available for all subjects treated with a BEAR Implant at each participating site. There is no control group.

ELIGIBILITY:
Inclusion Criteria for Prospective Cohort:

1. Scheduled to undergo ACL surgery with the BEAR Implant
2. Willing and able to provide informed consent
3. Willing and able to complete required follow-up visits and assessments

Inclusion Criteria for Retrospective Cohort:

1. Underwent ACL surgery with the BEAR Implant

Exclusion Criteria:

1. The subject is participating in another ACL trial or any other clinical trial where the study procedure or treatment might confound the study end point
2. Known allergy to bovine collagen, bovine gelatin or other bovine-derived products as contraindicated in the BEAR Implant labeling

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry will enroll consecutive subjects who meet the inclusion criteria with an expected sample size of up to 750 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation score at year 2 | 2 Years
  This is a survey patients complete about how their knee is feeling and functioning. Range is 0 to 100, with 100 indicating no problems and 0 indicating extreme problems.
Knee laxity based on the Lachman test at 1 year | 1 year
  The Lachman will be performed during physical exam.

SECONDARY OUTCOMES:
IKDC Subjective Knee Evaluation Score and Physical Exam at 6, 9 and 12 months post-surgery and according to standard of care | 6-12 months
  This is an examination performed of the knee. Scores are one of four measures: A (Normal), B (Nearly Normal), C (Abnormal) and D (Severely Abnormal). A is the best outcome and D is the worst.
Knee Injury and Osteoarthritis Outcome Score (KOOS) domains: Symptoms/Stiffness, Pain, Knee Related Quality of Life, and Knee Related Sports/Recreational Activities starting at 6, 9, 12 months and at 2 years after surgery | 6 months- 2 years post surgery
  This is a survey with 5 subscales (Pain, Symptoms, Function in Daily Living, Function in Sport and Recreation, and Knee Related Quality of Life). The range of each subscale is 0 to 100, with 100 indicating no problems and 0 indicating extreme problems. The subscales are reported individually and not combined.
Marx Activity Score at 6, 9, 12 months and at 2 years after surgery | 6 months thru 2 years
  Patients are asked to indicate approximately how many times in the past 12 months they performed each of these activities while at their healthiest and most active state. The four knee functions are rated on a 5-point scale of frequency and scores are added up to a maximum of 16 points with a higher score indicating more frequent participation.
Return to Sports Index (RSI) at 6, 9, 12 months and at 2 years after surgery | 6 months thru 2 years
  Measures the patients emotion, confidence, and risk appraisal when returning to sports after an ACL injury and/or reconstructive surgery. There are 12 questions and the subjects answer each in range is from 0 to 100. The response scale meaning is dictated by the question. The sum of all questions are reported, divided by 12,000 and multiplied by 100 to get a %.
VAS (Visual Analog Scale) Pain Score from post op through the first 12 months (approximately every 12 weeks) and at 2 years after surgery | 1 year
  A tool widely used to measure pain. The patient indicates his/her perceived pain intensity along a 100 mm horizontal line and this rate is then measure from the left edge to give a score.
Current Status Questionnaire | 2 years
  Elements include return to activity, pain medication use. No Score.
Pain Medication Use | 2 years
  Administered by questionnaire. No score.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Stanford, Redwood City, California
  - Steamboat Orthopaedic and Spine Institute, Steamboat Springs, Colorado
  - Advent Health, Orlando, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - Virtua Health, Marlton, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Victory Sports Medicine, Skaneateles, New York
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon

IPD SHARING:
Plan to Share IPD: No